CLINICAL TRIAL: NCT02531984
Title: Open Trial With Randomized Withdrawal of Treatment, to Evaluate the Efficacy of Azithromycin in the Treatment of Children With Non Cystic Fibrosis Bronchiectasis ( AZI-STOP Study )
Brief Title: The Efficacy of Azithromycin in Treating Children With Non Cystic Fibrosis Bronchiectasis
Acronym: AZI-STOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-26; RC12_3643 (Other: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Non Cystic Fibrosis Bronchiectasis in Children
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Withdrawal of Azithromycin treatment (Experimental)
  Interventions: Drug: Azithromycin
- ongoing Azithromycin treatment (Other)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
Bronchiectasis is characterized by a permanent and abnormal dilatation of a part of the bronchial tree. An accumulation of mucus in the respiratory tract ensues, resulting in frequent bacterial infections and eventual destruction of the lungs. Clinically, patients present with a chronic productive cough and episodes of acute respiratory exacerbations. Chronic respiratory failure can follow. Although its prevalence is largely unknown, bronchiectasis is considered to be a rare and orphan disease. There are numerous causes for this disease: sequelae of respiratory infections, immunodeficiency, genetic diseases like cystic fibrosis, primary ciliary dyskinesia….The focus of this study will be on non cystic fibrosis bronchiectasis in children.

Due to a lack of pediatric clinical trials, the management of children with this disease is widely based on the management of adults or patients with cystic fibrosis or pan-bronchiolitis. The treatment is based on respiratory physiotherapy, prevention of infections, administration of inhaled corticosteroids and anti biotherapy for acute exacerbations.

Recently, some studies have demonstrated the efficacy of a family of antibiotics, the macrolides, in the treatment of cystic fibrosis or pan-bronchiolitis in children. Indeed, taken 3 times a week during a long period of time, the macrolides, and specifically the azithromycin have shown some anti-inflammatory and tissue repairing properties, in addition to their antimicrobial properties.

Moreover, several studies conducted in the adult population have shown that the use of azithromycin has led to significant reduction in the frequency of respiratory exacerbations as well as an improvement in the quality of life.

The efficacy of azithromycin in these respiratory diseases has led to enlarge its use for the long term treatment of bronchiectasis. Yet, this type of treatment has no marketing authorization application.

No studies have been conducted in children, but individual examination of patients with bronchiectasis treated with azithromycin suggests an improvement of their symptoms.

Thus, the use of azithromycin in the treatment of bronchiectasis in children seems to be a promising therapy. However, its efficacy needs to be demonstrated by clinical trials led on a pediatric population with an adequate number of patients and a strong methodology in order to ensure validity and reliability of the results.

Therefore the investigators decided to conduct a comparative, prospective multicenter randomized study in this population.

This study intends to include 100 patients already treated by azithromycin for at least 6 months. After inclusion, they will be randomized in two groups of 50 patients each. The first group will continue the treatment and the other one will discontinue it.

The patients will be followed from the inclusion period (M0) until the onset of the first exacerbation for a maximum of 6 months (M6), with an intermediate health care visit after 3 months (M3).

In case of exacerbation, a health care visit will be scheduled; the patient will receive the appropriate treatment and he will be suspended from the study.

The duration of follow up for each patient is dictated by the occurrence of the first respiratory exacerbation, a maximum of 6 months .The total inclusion period is 12 months and the total duration of the study is 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with non cystic fibrosis bronchiectasis documented by chest CT scan , diagnosed since at least 2 years
* Already treated with azithromycin for at least 6 months
* Presented no respiratory exacerbation since one month
* Benefit from health insurance
* Have signed a consent (if appropriate age )
* Parents or legal guardian have given their written consent

Exclusion Criteria:

* Patients presenting a history of allergic reaction to azithromycin, érythromycine, another macrolide or Ketolide or an excipient of Zithromax
* Patients treated with dihydroergotamine or ergotamine , cisapride, colchicine
* Patients presenting severe hepatic failure
* Patients who are unlikely to adhere to the protocol and hence participate in the entire study ( as judged by the investigator )
* Patients who have not signed the protocol
* Patients whose parents are unable to understand the purpose and conditions of the study or are unable to give their consent.
* Patients already included in another clinical trial or are in an exclusion period from a previous clinical trial
* Patients whose ECG shows a QTc > 450 msec ( Zithromax is contraindicated )

Ages: 3 Years to 17 Years | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Time of onset of the first respiratory exacerbation in the two groups of patients: those who continued treatment with azithromycin and those who stopped the treatment | 6 months
  Exacerbations are defined by a combination of major and minor clinical criteria (Kapur et al, 2012) and the need for an antibiotic therapy for lower respiratory tract in case of acute infection. These criteria are evaluated by parents with the help of a daily diary; respiratory exacerbation is confirmed by a clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille